CLINICAL TRIAL: NCT03098160
Title: A Phase 1 Immunotherapy Study of Evofosfamide in Combination With Ipilimumab in Patients With Advanced Solid Malignancies
Brief Title: Immunotherapy Study of Evofosfamide in Combination With Ipilimumab
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Threshold Pharmaceuticals (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TH-CR-417
Record Dates: First submitted 2017-03-22; First posted 2017-03-31 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Pancreatic Cancer; Melanoma; Squamous Cell Carcinoma of the Head and Neck; Prostate Cancer
Keywords: Immunotherapy; Hypoxia; Evofosfamide; Ipilimumab; TH-302
MeSH Terms: conditions — Pancreatic Neoplasms; Melanoma; Squamous Cell Carcinoma of Head and Neck; Prostatic Neoplasms; Hypoxia | interventions — TH 302; Ipilimumab

STUDY DESIGN:
Intervention Model Description: During the initial phase of the study a maximum tolerated dose will be determined based on the dose escalation scheme in the protocol. Once this dose is established, enrollment will be expanded for each of the 4 disease cohorts at that dose level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evofosfamide plus Ipilimumab (Experimental): Ipilimumab to be administered at same dose. Evofosfamide dose to be determined during duration of trial
  Interventions: Drug: Evofosfamide; Drug: Ipilimumab

INTERVENTIONS:
Drug: Evofosfamide — Evofosfamide given on day one and in combination with Ipilimumab on day 8 of the first two cycles, Ipilimumab given alone on day 8 of last two cycles for a total of four 21 day dosing cycles.
Drug: Ipilimumab — Evofosfamide given on day one and in combination with Ipilimumab on day 8 of the first two cycles, Ipilimumab given alone on day 8 of last two cycles for a total of four 21 day dosing cycles.

SUMMARY:
An immunotherapy study combining ipilimumab and evofosfamide for the treatment of patients with confirmed metastatic or locally advanced prostate cancer, metastatic pancreatic cancer, melanoma or human papillomavirus (HPV) negative squamous cell carcinoma of head and neck that have failed to respond to standard therapy, progressed despite standard therapy, for which standard therapy does not offer the potential for increased survival.

DETAILED DESCRIPTION:
Tumor hypoxia can lead to poor effector T cell penetration and immunosuppressive signaling via myeloid-derived suppressor, myofibroblast and regulatory T cells. Disruption of these hypoxic regions within the tumor microenvironment by the hypoxia-directed cytotoxic agent evofosfamide may enhance the ability of the CTLA-4 checkpoint inhibitor ipilimumab to reject otherwise resistant solid tumors. Additionally, induction of immunogenic cell death of tumor cells by evofosfamide may enhance dendritic cell presentation of tumor antigens to lymphocytes in draining lymph nodes, leading to clonal expansion of tumor-specific T cells, especially in combination with ipilimumab.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be willing and able to review, understand, and provide written consent before study enrollment
2. Patients must have either a histologically-confirmed metastatic or locally advanced prostate cancer, metastatic pancreatic cancer, melanoma or human papillomavirus (HPV) negative squamous cell carcinoma of head and neck.
3. At least 18 years of age.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 (Karnofsky > 60 %)
5. Measurable disease as defined by irRECIST. Patients with castrate-resistant prostate cancer can have measurable or evaluable disease. Patients with evaluable disease must have documented evidence of progressive disease as defined by any of the following:

   1. Prostate-specific antigen (PSA) progression: minimum of 2 rising values (3 measurements) obtained a minimum of 7 days apart with the last result being at least >/= 1.0 ng/mL;
   2. New or increasing non-bone disease (RECIST 1.1 criteria);
   3. Positive bone scan with 2 or more new lesions (PCWG3)
6. Adequate bone marrow function within 7 days and defined as:

   1. White Blood Cell (WBC) ≥ 2500 cells/mm3
   2. Absolute neutrophil count (ANC) ≥ 1,500 cells/mm3cells
   3. Absolute lymphocyte count (ALC) >1000 cells/mm3
   4. Hemoglobin ≥ 9 g/dL
   5. Platelets (PLT) ≥ 75,000 cells/mm3
7. Acceptable renal function within 7 days defined as serum creatinine ≤ 2.0 times the institutional upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 mL/min (by the Cockcroft Gault formula).
8. Acceptable liver function within 7 days of day 1 of therapy defined as:

   1. • Bilirubin ≤ 1.5 times institutional ULN; does not apply to patients diagnosed with Gilbert's syndrome.
   2. • AST (SGOT) and ALT (SGPT) ≤ 3 times institutional ULN; if liver metastases are present, then ≤ 5 times ULN is allowed.
9. QTc interval of ≤ 450 msec (males) or 470 msec (females) calculated according to Fridericia's formula (QTc = QT/RR0.33; RR=RR interval)
10. Ability and availability to complete all prescribed biopsies (prior to the first evofosfamide dose and between day 15 of Cycle 2 and day 8 of Cycle 3)
11. At least 3 weeks from previous cytotoxic chemotherapy or radiation therapy and at least 5 half-lives or 6 weeks, whichever is shorter, after targeted or biologic therapy excepting prior treatment with CTLA 4, PD-1, or PD-L1 blocking antibodies for which only a 2 week interval is required. Patients with prostate cancer, unless orchiectomy has been performed in them, may continue to receive androgen deprivation therapy (ADT), anti-androgen therapy or therapy that interferes with androgenic stimulation.
12. Patients must have recovered from toxicity related to prior therapy to at least grade 1 (defined by CTCAE 4.0) or baseline level. Chronic stable grade 2 peripheral neuropathy secondary to neurotoxicity from prior therapies may be considered on a case by case basis by the Principal Investigator.
13. Female patients of childbearing age must have a negative serum HCG test within 7 days of study enrollment, unless prior hysterectomy or menopause (defined as age ≥ 55 years and twelve consecutive months without menstrual activity). Female patients should not become pregnant or breast-feed while on this study.
14. Sexually active male and female patients should use effective birth control (abstinence; hormonal or barrier method) for the duration of the study and at least 2 months from last dose.

Exclusion Criteria:

1. Active/uncontrolled autoimmune disease: patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis [scleroderma], Systemic Lupus Erythematosus or autoimmune vasculitis [e.g., Wegener's Granulomatosis] are excluded from this study.
2. Patients with history of any Grade 3 or Grade 4 adverse events from prior ipilimumab therapy, if administered in the past.
3. Patients with history of mild autoimmune disorders - including but not limited to - mild psoriasis or Hashimoto's hypothyroidism, may be included at the discretion of the principle investigator.
4. History of acute diverticulitis, intra-abdominal abscess, GI obstruction, abdominal carcinomatosis or other known risk factors for bowel perforation.
5. Patients on long term systemic steroids (>10 mg daily prednisone equivalent). Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune thyroiditis only requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger are permitted to enroll at the discretion of the principle investigator. Inhaled or topical steroids are permitted in the absence of active autoimmune disease.
6. Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of AEs: e.g. a condition associated with frequent diarrhea or chronic skin conditions, recent surgery or colonic biopsy from which the patient has not recovered, or partial endocrine organ deficiencies.
7. Receiving QT-prolonging drugs with a risk of causing torsades de pointes (See Appendix E), unless ECG meets inclusion criteria on a stable dose of the drug and with discussion and agreement with the project clinician
8. History of risk factors for TdP, including family history of long QT syndrome.
9. Sustained systolic blood pressure (BP) >140 mm Hg or <90 mm Hg, diastolic BP >100 mm Hg or <60 mm Hg
10. Patients with newly diagnosed, uncontrolled and or untreated cancer; related central nervous system diseases are excluded.
11. Uncontrolled intercurrent illness, including, but not limited to, myocardial infarction within 6 months, unstable symptomatic ischemic heart disease, active uncontrolled infection requiring systemic therapy, or psychiatric illness/social situations that would limit compliance with study requirements.
12. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days of day 1 of therapy.
13. Current evidence of active and uncontrolled infection, NYHA Class III-IV CHF, documented Child's class B and C cirrhosis, active pancreatitis or uncontrolled medical disease which in the opinion of the investigator could compromise assessment of efficacy.
14. Known human immunodeficiency virus (HIV)-positive unless on highly active antiretroviral therapy (HAART), and/or known Hepatitis B or C on treatment. Drug interactions between those agents and these experimental agents are wholly unknown (screening not required).
15. Known hypersensitivity to the components of study drugs, its analogs, or drugs of similar chemical or biologic composition.
16. Any live vaccine or non-oncology vaccine therapy used for prevention of infectious diseases (for up to one month prior to or after any dose of ipilimumab).
17. Concomitant therapy with any of the following: IL-2, interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; or other investigational therapies.
18. Receiving medications that are strong inhibitors or inducers of CYP3A4 (Appendix D).
19. Use of any other concurrent investigational agents or anticancer agents including hormonal therapy, except in the case of prostate cancer patients who are being treated anti-androgen or bone targeting therapies.
20. Female patients who have been on hormone replacement therapy (HRT) for menopausal symptoms for a period of at least 2 months will not be excluded from the study provided the HRT regimen remains unchanged during the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) determined after maximally tolerated dose is set and four dose expansion cohorts have evaluable data | Approximately 8-12 months
  Threshold and MD Anderson Cancer Center to evaluate patient safety data to determine proper dose

SECONDARY OUTCOMES:
Maximum tolerated dose (MTD) of this therapy based on number of dose limiting toxicities that occur during the dose escalation phase | Approximately 4-6 months
  Threshold and MD Anderson Cancer Center to evaluate patient safety data to determine proper dose
Number of participants with treatment related adverse events | Approximately 2 years
  Safety grading based on CTCAE guidelines
Change from tumor diameter baseline | Approximately 2 years
  Antitumor efficacy based on irRECIST

CONTACTS AND LOCATIONS:
Overall Officials: David Hong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Safety and efficacy data may be shared in the form of a paper or trials in progress poster at a conference. Additionally, data may be shared via the clinical study report.